CLINICAL TRIAL: NCT06042166
Title: A Postpartum Adaptation Study of the Connecting and Reflecting Experience Parenting Program
Acronym: PMAD-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: American Psychological Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2023-15124
Record Dates: First submitted 2023-09-06; First posted 2023-09-18 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Postpartum Depression; Postpartum Anxiety; Parenting Stress; Parent Child Relationships
Keywords: postpartum depression; group therapy; parenting stress; short-term therapy; parenting support; postpartum anxiety; perinatal mood and anxiety disorders; mentalizing; parental reflective functioning; attachment
MeSH Terms: conditions — Depression, Postpartum; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Connecting and Reflecting Experience (CARE) Program (Experimental): Participants will enroll in a 12-session CARE parenting group therapy.
  Interventions: Behavioral: Connecting and Reflecting Experience (CARE) Program

INTERVENTIONS:
Behavioral: Connecting and Reflecting Experience (CARE) Program — The intervention consists of a 12-session mentalizing-focused parenting group, which will involve weekly one-hour telehealth therapy sessions with up to 7 postpartum parents per group and 1 to 2 facilitators. CARE is a therapy focused on parents' reflective capacity, or the ability to consider how our own and our children's thoughts, feelings, intentions, and other mental states shape behavior and parent-child relationships.

SUMMARY:
Experiencing postpartum mood and/or anxiety disorders (like postpartum depression; PMADs) can make parenting challenging, but group therapy may help both these parents and their babies. This study will test whether postpartum parents with PMADs find a 12-session parenting group therapy to be likable, doable, and helpful for mental health, parenting stress, and relationship with their infant. The therapy that is being tested is called the Connecting and Reflecting Experience (CARE) parenting program, which has not yet been used specifically with postpartum parents with PMADs, but has been found to be appealing and helpful among parents/caregivers of older children with mental health conditions. CARE focuses on parents' ability to consider how their own and their children's thoughts, feelings, intentions, and other mental states shape behavior and parent-child relationships. Participants in the study will be asked to fill out surveys before, during, and after participating in the group therapy. Adults may be eligible to participate in the study if they gave birth to an infant who is now 3 to 12 months old, are receiving postpartum medical and/or mental health care at Montefiore Medical Center, and have experienced postpartum depression and/or anxiety.

ELIGIBILITY:
Inclusion Criteria:

* Birthing parent (of any gender) of an infant age 3-12 months old at time of enrollment
* Receiving postpartum OB/GYN or mental health services at Montefiore Medical Center
* Experienced or currently experiencing moderate to high levels of depression and/or anxiety symptoms in the postpartum period
* English-speaking

Exclusion Criteria:

* Prior participation in a Connecting and Reflecting Experience (CARE) group at any time
* Participation in another parenting-focused group during the current postpartum period
* Current episode of psychosis or mania or active suicidal ideation
* Serious psychiatric, neurocognitive, or substance use related difficulties necessitating a higher level of care than outpatient support (e.g., current inpatient treatment) or that, in the judgment of the PI, would impede group participation (e.g., severe cognitive impairment)

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-08-16 (Actual); Primary Completion 2025-11-11 (Actual); Study Completion 2025-11-11 (Actual)

PRIMARY OUTCOMES:
Change from Baseline to Post-Treatment in Postpartum Anxiety Score | The BAI will be administered at baseline (approximately 0-2 weeks pre-treatment) and at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in postpartum anxiety will be measured using the total score on a self-reported questionnaire: the 21-item Beck Anxiety Inventory (BAI; Beck et al, 1988). Total scores range from 0 to 63, with higher scores indicating higher anxiety symptoms.
Change from Baseline to Post-Treatment in Postpartum Depression Score | The EPDS will be administered at baseline (approximately 0-2 weeks pre-treatment) and at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in postpartum depression will be measured using the total score on a self-reported questionnaire: the Edinburgh Postnatal Depression Scale (EPDS; Cox, Holden, & Sagovsky, 1987). Total scores range from 0 to 30, with higher scores indicating higher depression symptoms.
Change from Baseline to Post-Treatment in Parenting Stress Score | The PSI-SF will be administered at baseline (approximately 0-2 weeks pre-treatment) and at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in parenting stress will be measured using the total score on a self-reported questionnaire: the 36-item Parenting Stress Index, Short-Form (PSI-SF; Abidin, 2012). Total scores range from 36 to 180. Raw scores can be converted to percentile based on a normed sample. Higher raw and percentile scores indicate higher levels of parenting stress. Scores falling between the 16th and 84th percentiles are considered within the normal range of parenting stress, scores between the 85th and 89th percentiles are considered high, and scores at the 90th percentile and above are considered in the clinically significant range.
Change from Baseline to Post-Treatment in Parental Reflective Functioning | The PRFQ will be administered at baseline (approximately 0-2 weeks pre-treatment) and at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in parental reflective functioning will be measured using subscale scores on a self-reported questionnaire: the 18-item Parental Reflective Functioning Questionnaire (PRFQ; Luyten et al., 2017). The PRFQ has three subscales, each of which has a score range from 6 to 42. Though threshold scores have not been established for the PRFQ, "adaptive" subscale scores would be in the mid-range for Certainty about Mental States, low range for Prementalizing Modes, and high range for Interest and Curiosity about Mental States.
Change from Baseline to Post-Treatment in Parent-Infant Bonding | The PBQ will be administered at baseline (approximately 0-2 weeks pre-treatment) and at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in parent-infant bonding will be measured using subscale scores on a self-reported questionnaire: the 25-item Postpartum Bonding Questionnaire (PBQ; Brockington et al., 2001). The PBQ has 4 subscales. Scale 1 (12 items) has a score range from 0 to 60; scores above 12 are considered "high" in impaired bonding. Scale 2 (7 items) has a score range from 0 to 35; scores above 17 are considered "high" in relational rejection/anger. Scale 3 (4 items) has a score range from 0 to 20; scores above 10 are considered "high" in anxiety about infant care. Scale 4 (2 items) has a range from 0 to 10; scores above 3 are considered "high" in aggression risk.
Post-treatment rating of treatment acceptability and feasibility | This survey will be administered at post-treatment (i.e., after completion of Session 12, approximately 15 weeks after baseline measurement).
  Participants will complete a brief self-reported survey developed for this study to assess their perceptions of treatment acceptability and feasibility. Participants will rate their sense of satisfaction, enjoyment, helpfulness, and comfort with the CARE group program on a scale from 0 to 10, where higher scores indicate greater treatment acceptability. Participants will also rate how challenging aspects of group were (i.e., attendance and emotional content) from 0 to 10, where higher scores indicate lower program feasibility/greater challenge. Participants will also be asked to provide qualitative feedback regarding their impressions of the program.
Change from Session 1 to Session 12 in Therapeutic Group Processes | The TFI-19 will be administered after participants complete Session 1 of group (approximately 0-2 weeks after baseline measurement) and again at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in therapeutic group processes will be measured using subscales on a self-reported questionnaire: the revised Therapeutic Factors Inventory-19 item version (TFI-19; Joyce et al., 2011). Each item is scored from 1 to 7. Subscale scores are generated as an average/mean of item ratings. Higher subscale scores indicate greater perceptions of indicated therapeutic factors within their CARE group: Instillation of Hope (4 items), Secure Emotional Expression (7 items), Awareness of Relational Impact (5 items), and Social Learning (3 items).

SECONDARY OUTCOMES:
Change from Baseline to Post-Treatment in Infant Temperament | The IBQ-VSF will be administered at baseline (approximately 0-2 weeks pre-treatment) and at post-treatment (after completion of Session 12, approximately 15 weeks after baseline measurement).
  Change in infant temperament will be measured using a parent-reported questionnaire: the 37-item Infant Behavior Questionnaire, Revised, Very Short Form (IBQ-VSF; Putnam et al., 2014). The IBQ-VSF has 3 subscales for which mean scores ranging from 1 to 7 are generated. The Surgency subscale has 13 items; higher scores indicate greater infant emotional surgency. The Negative Affect subscale has 12 items; higher scores indicate greater infant negative affect. The Effortful Control subscale has 12 items; higher scores indicate greater infant effortful control.

CONTACTS AND LOCATIONS:
Overall Officials: Amanda Zayde, Psy.D., Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

IPD SHARING:
Plan to Share IPD: No
The study is a small pilot and thus data sharing is not appropriate at this stage.

REFERENCES:
- [Background] Zayde A, Kilbride A, Kucer A, Willis HA, Nikitiades A, Alpert J, Gabbay V. Connection During COVID-19: Pilot Study of a Telehealth Group Parenting Intervention. Am J Psychother. 2022 Jun 15;75(2):67-74. doi: 10.1176/appi.psychotherapy.20210005. Epub 2021 Sep 16. PMID 34525847
- [Background] Zayde A, Derella OJ, Kilbride A. Safe haven in adolescence: Improving parental reflective functioning and youth attachment and mental health with the Connecting and Reflecting Experience. Infant Ment Health J. 2023 Mar;44(2):268-283. doi: 10.1002/imhj.22042. Epub 2023 Mar 2. PMID 36862314
- [Background] Zayde A, Prout TA, Kilbride A, Kufferath-Lin T. The Connecting and Reflecting Experience (CARE): theoretical foundation and development of mentalizing-focused parenting groups. Attach Hum Dev. 2021 Jun;23(3):293-309. doi: 10.1080/14616734.2020.1729213. Epub 2020 Feb 19. PMID 32072881
- [Background] Putnam SP, Helbig AL, Gartstein MA, Rothbart MK, Leerkes E. Development and assessment of short and very short forms of the infant behavior questionnaire-revised. J Pers Assess. 2014;96(4):445-58. doi: 10.1080/00223891.2013.841171. Epub 2013 Nov 9. PMID 24206185
- [Background] Luyten P, Mayes LC, Nijssens L, Fonagy P. The parental reflective functioning questionnaire: Development and preliminary validation. PLoS One. 2017 May 4;12(5):e0176218. doi: 10.1371/journal.pone.0176218. eCollection 2017. PMID 28472162
- [Background] Goodman JH, Santangelo G. Group treatment for postpartum depression: a systematic review. Arch Womens Ment Health. 2011 Aug;14(4):277-93. doi: 10.1007/s00737-011-0225-3. Epub 2011 Jul 1. PMID 21720793
- [Background] Brockington IF, Oates J, George S, Turner D, Vostanis P, Sullivan M, Loh C, Murdoch C. A screening questionnaire for mother-infant bonding disorders. Archives of Women's Mental Health. 2001; 3: 133-140.
- [Background] Beck, AT, Steer, RA. Beck Anxiety Inventory Manual. San Antonio, TX: Psychological Corporation. 1993.
- [Background] Abidin, R. R. (2012). Parenting Stress Index (4th ed.). Lutz, FL: PAR.
- [Background] Cox JL, Holden JM, Sagovsky R. Detection of postnatal depression. Development of the 10-item Edinburgh Postnatal Depression Scale. Br J Psychiatry. 1987 Jun;150:782-6. doi: 10.1192/bjp.150.6.782. PMID 3651732
- [Background] Joyce AS, MacNair-Semands R, Tasca GA, Ogrodniczuk JS. Factor structure and validity of the Therapeutic Factors Inventory-Short Form. Group Dynamics. 2011; 15(3): 201-219.